CLINICAL TRIAL: NCT02244177
Title: Relationship of Essential Hypertension and Its Treatments on the Postoperative Pain Management: a Prospective, Observational, Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Yuan-Yi Chia, anesthesia doctor, Kaohsiung Veterans General Hospital.
Other Study IDs: VGHKS-103-080
Record Dates: First submitted 2014-09-10; First posted 2014-09-18 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- normotension group: Until 11,March, 2015, 31 cases are collected.
- hypertension group without treatment: Until 11,March, 2015, 60 cases are collected.
- hypertension group with antihypertensive treatment: (ACEI, beta-blocker, Ca blocker, Diuretics) prior to the surgery.
  Until 11,March, 2015, 59 cases are collected.

SUMMARY:
Numbers of postoperative PCA related side effects among three groups will be determined by comparing and analyzing frequency distributions. To determine whether the patients with hypertension require less post operative opiate analgesics than others, multivariate analysis with repeated measures will be performed to identify the major and the minor factors predicting the use of postoperative pain therapy. The major aim of the study is to test the hypothesis that the morphine comsumpted by the hypertension group is less than those of the normotension group. The minor aims for the study are the difference related to pain intensity, or the incidence of side effects among groups.

ELIGIBILITY:
Inclusion Criteria:

* 300 eligible subjects
* No contraindication for inhalation anesthesia
* Elective surgery
* Age between 20-75 y/o
* No contraindication for postoperative morphine pain control
* Female or male
* Essential hypertension stage I and II (140<=SBP<=180; 90<=DBP<=110)

Exclusion Criteria:

* Liver disease
* Renal disease
* Those who is presumed to go to ICU after surgery
* The patients with dementia or conscious disturbance
* Pregnancy or breast feeding
* Secondary hypertension
* events in recent 6 months myocardial infarction cardiac bypass surgery unstable angina cerebrovascular events congestive heart failure significant arrhythmia thoracic surgery

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those patients enrolled will be divided into three groups as follows As the treatment and choice of drugs for hypertension is complex but internation guideline-oriented. We would like to enroll enough sample size in the hypertensive groups and subgroups.
  1. Normaltension group (control group)
  2. Hypertension without treatment
  3. Hypertension with treatment as follows (according to subject's daily routine Tx, the PI not involved into the choice and further manitence of drugs) I. Hypertension with treatment with ACEI II. Hypertension with treatment with β blocker III. Hypertension with treatment with Ca channel blocker IV. Hypertension with treatment with diuretics
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Pain | Post-operation Day1 to Day4

SECONDARY OUTCOMES:
Morphine consumption | Post-operation Day1 to Day4

OTHER OUTCOMES:
side effects | Post-operation Day1 to Day4

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan